CLINICAL TRIAL: NCT03071133
Title: Asunaprevir/Daclatasvir/Beclabuvir Fixed-Dose Combination Safety Surveillance in Japanese Patients With Chronic Hepatitis C (HCV) or Japanese Patients With Compensated Cirrhosis
Brief Title: Real-world Incidence Proportion of Hepatic Toxicity and All Adverse Drug Reactions (ADRs) in Japanese Patients Receiving Daclatasvir (DCV) Trio Therapy
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI443-144
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An observational, postmarketing commitment following the marketing authorization for DCV Trio therapy in Japan

ELIGIBILITY:
Inclusion Criteria:

* Patients who are initiating the treatment with DCV Trio therapy under the approved indications, dosage, and administration

Exclusion Criteria:

* Patients who use the DCV Trio off label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Japan who are initiating treatment with DCV Trio therapy
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Aspartate Aminotransferase (AST) elevation | Up to 36 weeks
  measured by immunoassay
Incidence of Alanine Aminotransferase (ALT) elevation | Up to 36 weeks
  measured by immunoassay
Incidence of Total Bilirubin (tBili) elevation | Up to 36 weeks
  measured by immunoassay

SECONDARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) in HCV patients treated with DCV Trio therapy in Japan | Up to 36 weeks
  measured by adverse events
Proportion of patients with undetectable HCV RNA at 12 weeks post-treatment (SVR12) | Up to 24 weeks
  measured by number of patients
Proportion of patients with undetectable HCV RNA at 24 weeks post-treatment (SVR24) | Up to 36 weeks
  measured by number of patients
Percentage of patients to experience virologic breakthrough | Up to 36 weeks
  measured by percentage of patients

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm